CLINICAL TRIAL: NCT03519386
Title: Prospective, Randomized Phase III Study Comparing Two Models of a Travoprost Intraocular Implant to Timolol Maleate Ophthalmic Solution, 0.5%
Brief Title: Randomized Study Comparing Two Models of a Travoprost Intraocular Implant to Timolol Maleate Ophthalmic Solution, 0.5%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC-010
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Implant Group 1 (Experimental): G2-TR intraocular implant containing travoprost 75 mcg with high elution rate, plus postoperative placebo eye drops.
  Interventions: Combination Product: G2-TR intraocular implant containing travoprost
- Implant Group 2 (Experimental): G2-TR intraocular implant containing travoprost 75 mcg with low elution rate, plus postoperative placebo eye drops.
  Interventions: Combination Product: G2-TR intraocular implant containing travoprost
- Control Group (Active Comparator): Sham surgery + active-comparator eye drops
  Interventions: Drug: Sham surgery + active-comparator eye drops

INTERVENTIONS:
Combination Product: G2-TR intraocular implant containing travoprost — Provided in Arm/Group descriptions.
  Other Names: Implant Group
  Arms: Implant Group 1; Implant Group 2
Drug: Sham surgery + active-comparator eye drops — Sham surgery plus postoperative active-comparator eye drops (timolol maleate ophthalmic solution, 0.5%).
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
Phase III study to compare the safety and efficacy of intraocular implants containing travoprost at two different elution rates versus Timolol Maleate Ophthalmic Solution, 0.5% (timolol) in reducing elevated intraocular pressure in subjects with open-angle glaucoma (OAG) or ocular hypertension (OHT).

DETAILED DESCRIPTION:
This is a prospective, randomized, double-masked, active-controlled, parallel-group, multi-center trial comparing the efficacy and safety of the Model G2TR 063 Travoprost Intraocular Implant and the Model G2TR-125 Travoprost Intraocular Implant to topical timolol in subjects with OAG or OHT. The staff who record key efficacy measures and the study subjects will remain masked to study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open-angle glaucoma or ocular hypertension.
* C/D ratio ≤ 0.8
* Zero to three preoperative ocular hypotensive medications

Exclusion Criteria:

* Active corneal inflammation or edema.
* Retinal disorders not associated with glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Stephens, O.D., Study Chair — Glaukos Corporation
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

REFERENCES:
- [Derived] Singh IP, Berdahl JP, Sarkisian SR Jr, Voskanyan LA, Ang RE, Doan LV, Applegate D, Shen Y, Katz LJ, Kothe AC, Navratil T. Long-Term Safety and Efficacy Evaluation of Travoprost Intracameral Implant Based on Pooled Analyses from Two Phase III Trials. Drugs. 2024 Oct;84(10):1299-1311. doi: 10.1007/s40265-024-02074-9. Epub 2024 Sep 6. PMID 39240530
- [Derived] Bacharach J, Doan LV, Stephens KG, Usner DW, Kothe AC, Katz LJ, Navratil T. Travoprost Intracameral Implant Demonstrates Superior IOP Lowering Versus Topical Prostaglandin Analog Monotherapy in Patients with Open-Angle Glaucoma or Ocular Hypertension. Ophthalmol Ther. 2024 Sep;13(9):2357-2367. doi: 10.1007/s40123-024-00992-1. Epub 2024 Jul 10. PMID 38985408
- [Derived] Sarkisian SR, Ang RE, Lee AM, Berdahl JP, Heersink SB, Burden JH, Doan LV, Stephens KG, Applegate D, Kothe AC, Usner DW, Katz LJ, Navratil T. Travoprost Intracameral Implant for Open-Angle Glaucoma or Ocular Hypertension: 12-Month Results of a Randomized, Double-Masked Trial. Ophthalmol Ther. 2024 Apr;13(4):995-1014. doi: 10.1007/s40123-024-00898-y. Epub 2024 Feb 12. PMID 38345710
- [Derived] Belamkar A, Harris A, Zukerman R, Siesky B, Oddone F, Verticchio Vercellin A, Ciulla TA. Sustained release glaucoma therapies: Novel modalities for overcoming key treatment barriers associated with topical medications. Ann Med. 2022 Dec;54(1):343-358. doi: 10.1080/07853890.2021.1955146. PMID 35076329

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: subjects required to undergo washout of prior IOP-lowering medication(s) if applicable and to meet inclusion/exclusion criteria
Period: Overall Study
Arm/Group | Implant Group 1 | Implant Group 2 | Control Group
Started | 200 | 197 | 193
Month 3 | 196 | 195 | 189
Month 12 | 190 | 192 | 183
Completed | 0 | 0 | 0
Not Completed | 200 | 197 | 193
Not completed — Withdrawal by Subject | 4 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Death | 1 | 0 | 4
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Explanted | 2 | 1 | 0
Not completed — Ongoing in study | 190 | 192 | 183

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Implant Group 1 | Implant Group 2 | Control Group | Total
Number analyzed (Participants) | 200 | 197 | 193 | 590
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 102 | 91 | 93 | 286
  >=65 years | 98 | 106 | 100 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.5) | 63.2 (12.6) | 63.8 (11.4) | 63.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 99 | 108 | 316
  Male | 91 | 98 | 85 | 274
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 15 | 10 | 34
  Not Hispanic or Latino | 191 | 179 | 180 | 550
  Unknown or Not Reported | 0 | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 15 | 19 | 16 | 50
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 38 | 50 | 41 | 129
  White | 143 | 120 | 128 | 391
  More than one race | 3 | 7 | 5 | 15
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 186 | 183 | 179 | 548
  Philippines | 14 | 14 | 14 | 42
Baseline Mean Diurnal IOP [Mean (Standard Deviation); unit: mmHg] — Average of the intraocular pressure at the 8AM, 10AM and 4PM timepoints following washout from prior IOP-lowering medication(s), if applicable
  mmHg | 24.2 (2.78) | 24.0 (2.81) | 24.1 (2.68) | 24.1 (2.76)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Diurnal IOP (as Measured at 8AM and 10AM) Through 3 Months Postoperative
Description: Change from time-matched baseline in IOP at 8AM and 10AM at Day 10, Week 6 and Month 3.
  Day 10 8AM IOP minus Baseline 8AM IOP; Day 10 10AM IOP minus Baseline 10AM IOP; Week 6 8AM IOP minus Baseline 8AM IOP; Week 6 10AM IOP minus Baseline 10AM IOP; Month 3 8AM IOP minus Baseline 8AM IOP; Month 3 10AM IOP minus Baseline 10AM IOP.
Time Frame: 3 months
Population: intent to treatment analysis set which includes all randomized subjects with analyses performed according to original treatment assignment, regardless of actual treatment received
Measure: Least Squares Mean (Standard Error); unit: mmHg
Units Other Than Participants: study eyes
Arm/Group | Implant Group 1 | Implant Group 2 | Control Group
Number analyzed (Participants) | 200 | 197 | 193
Number analyzed (study eyes) | 200 | 197 | 193
mmHg
  Day 10, 8AM | -8.40 (0.24) | -8.48 (0.24) | -7.69 (0.24)
  Day 10, 10AM | -8.35 (0.24) | -8.44 (0.24) | -7.20 (0.24)
  Week 6, 8AM | -7.34 (0.24) | -7.26 (0.25) | -7.09 (0.25)
  Week 6, 10AM | -7.59 (0.24) | -7.62 (0.24) | -6.85 (0.24)
  Month 3, 8AM | -6.59 (0.26) | -6.59 (0.26) | -6.69 (0.27)
  Month 3, 10AM | -6.56 (0.26) | -6.68 (0.26) | -6.52 (0.27)
Statistical Analysis 1: Comparison: Implant Group 2 vs Control Group; Day 10, 8AM Difference between Implant Group 2 and timolol; Test type: Non-Inferiority — criteria for statistical and clinical non-inferiority: upper limit of the 95% CI of the difference between the implant group and the timolol group was < 1.5 mmHg and also < 1 mmHg for all 6 timepoints for Implant Group 2 vs. Timolol; Fixed sequence hierarchical testing procedure was used, first testing for non-inferiority of Implant Group 2 to timolol at all 6 timepoints before testing non-inferiority of Implant Group 1 to timolol; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-1.45 to -0.13]
Statistical Analysis 2: Comparison: Implant Group 2 vs Control Group; Day 10, 10AM Difference between Implant Group 2 and timolol; Test type: Non-Inferiority — criteria for statistical and clinical non-inferiority: upper limit of the 95% CI of the difference between the implant group and the timolol group was < 1.5 mmHg and also < 1 mmHg for all 6 timepoints for Implant Group 2 vs Timolol; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.24, 95% CI 2-sided [-1.92 to -0.56]
Statistical Analysis 3: Comparison: Implant Group 2 vs Control Group; Week 6, 8AM Difference between Implant Group 2 and timolol; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.86 to 0.51]
Statistical Analysis 4: Comparison: Implant Group 2 vs Control Group; Week 6, 10AM Difference between Implant Group 2 and timolol; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.43 to -0.11]
Statistical Analysis 5: Comparison: Implant Group 2 vs Control Group; Month 3, 8AM Difference between Implant Group 2 and timolol; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.63 to 0.82]
Statistical Analysis 6: Comparison: Implant Group 2 vs Control Group; Month 3, 10AM Difference between Implant Group 2 and timolol; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.89 to 0.57]
Statistical Analysis 7: Comparison: Implant Group 1 vs Control Group; Day 10, 8AM Difference between Implant Group 1 vs. Timolol; Test type: Non-Inferiority — criteria for statistical and clinical non-inferiority: upper limit of the 95% CI of the difference between the implant group and the timolol group was < 1.5 mmHg and also < 1 mmHg for all 6 timepoints for Implant Group 1 vs. Timolol; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.72, 95% CI 2-sided [-1.38 to -0.06]
Statistical Analysis 8: Comparison: Implant Group 1 vs Control Group; Day 10, 10AM Difference between Implant Group 1 vs. Timolol; Test type: Non-Inferiority — criteria for statistical and clinical non-inferiority: upper limit of the 95% CI of the difference between the implant group and the timolol group was < 1.5 mmHg and also < 1 mmHg for all 6 timepoints for Implant Group 1 vs Timolol; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-1.83 to -0.48]
Statistical Analysis 9: Comparison: Implant Group 1 vs Control Group; Week 6, 8AM Difference between Implant Group 1 and timolol; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 7]; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.93 to 0.43]
Statistical Analysis 10: Comparison: Implant Group 1 vs Control Group; Week 6, 10AM Difference between Implant Group 1 and timolol; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 8]; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.40 to -0.08]
Statistical Analysis 11: Comparison: Implant Group 1 vs Control Group; Month 3, 8AM Difference between Implant Group 1 and timolol; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 7]; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.62 to 0.83]
Statistical Analysis 12: Comparison: Implant Group 1 vs Control Group; Month 3, 10AM Difference between Implant Group 1 and timolol; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 8]; [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.77 to 0.69]

2. Secondary Outcome: Mean IOP (Control Group vs. Each Implant Group) Through 12 Months Postoperative
Description: Difference in mean IOP, between each test group and the control group, for IOP measurements through the Month 12 follow-up visit
Time Frame: 12 months
Reporting Status: Not Posted, anticipated posting 2025-06

ADVERSE EVENTS:
Time Frame: 12 months post-operative
Description: The safety analysis set includes all subjects who were randomized & received >= 1 dose of study treatment, with subjects grouped according to their actual treatment received. 1 subject was randomized & not treated, & 4 subjects received treatment that differed from their randomization assignment: 1 randomized to Group 1 was treated with Control; 1 randomized to Control was treated as Group 1; 1 randomized to Group 2 was treated with Control; and 1 randomized to Group 2 was treated as Group 1.
Arm/Group | Implant Group 1 | Implant Group 2 | Control Group
All-Cause Mortality (participants affected / at risk) | 2/200 | 0/195 | 4/194
Serious Adverse Events (participants affected / at risk) | 5/200 | 6/195 | 7/194
Other Adverse Events (participants affected / at risk) | 16/200 | 21/195 | 4/194
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant Group 1 (N=200) | Implant Group 2 (N=195) | Control Group (N=194)
Combined adverse events in Cardiac Disorders SOC (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2) — All AEs in SOC combined to prevent unmasking in this ongoing double-masked trial
Combined adverse events in Musculoskeletal and Connective Tissue Disorders SOC (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) — All AEs in SOC combined to prevent unmasking in this ongoing double-masked trial
Combined adverse events in Infections and Infestations SOC (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) — All AEs in SOC combined to prevent unmasking in this ongoing double-masked trial
Combined adverse events in Psychiatric Disorders SOC (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) — All AEs in SOC combined to prevent unmasking in this ongoing double-masked trial
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant Group 1 (N=200) | Implant Group 2 (N=195) | Control Group (N=194)
iritis (Eye disorders) | 1 (1) | 12 (12) | 0 (0)
intraocular pressure increased (Investigations) | 15 (15) | 9 (9) | 4 (4)

LIMITATIONS AND CAVEATS:
This is an ongoing double-masked trial. Therefore, limited adverse event data are presented in order to prevent unmasking.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of data from this study.

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03519386/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03519386/SAP_001.pdf